CLINICAL TRIAL: NCT03478033
Title: The Efficacy and Safety Evaluation of Standardized Treatment Included Rifampicin or Rifabutin in HIV/AIDs Patients Combined With Pulmonary Tuberculosis. A Prospective Study.
Brief Title: Rifampicin vs Rifabutin in HIV/AIDS Patients Combined With Tuberculosis
Acronym: RRHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Collaborators: The Guangxi Zhuang Autonomous Region Longtan hospital (Unknown); The Fourth People's Hospital of Nanning (Other); Shenzhen Third People's Hospital (Other); Yunnan Provincial Infectious Disease Hospital (Other); Zhejiang University (Other); Chongqing Public Health Medical Center (Other)
Responsible Party: Principal Investigator, Hongzhou Lu, vice director, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017ZX10202101-002
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Tuberculosis, Pulmonary; AIDS
Keywords: Tuberculosis; AIDS; Rifampicin; Rifabutin
MeSH Terms: conditions — Tuberculosis, Pulmonary; Acquired Immunodeficiency Syndrome; Tuberculosis | interventions — Rifampin; Rifabutin

STUDY DESIGN:
Intervention Model Description: Participates are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifampicin group (Active Comparator): Rifampicin group: Intensive treatment（4 types of anti-TB medicines）for 2 months, then isoniazid and rifampicin for 4 months of consolidation therapy.
  isoniazid: 10-15mg/kg rifampicin: 10-20mg/kg pyrazinamide: 30-40mg/kg thambutol: 0.75(W<50kg)；1.0 g/d（W≥50kg）
  Interventions: Drug: Rifampicin
- Rifabutin group (Experimental): Rifabutin group: Intensive treatment（4 types anti-TB medicines）for 2 months,then isoniazid and rifabutin for 4 months of consolidation therapy.
  isoniazid: 10-15mg/kg rifabutin: 0.45g/d(W<50kg); 0.6g/d( W≥50kg） pyrazinamide: 30-40mg/kg thambutol: 0.75(W<50kg)；1.0 g/d（W≥50kg）
  Interventions: Drug: Rifabutin

INTERVENTIONS:
Drug: Rifampicin — Rifampicin capsules, 150mg
  Other Names: Rifampicin/INH/EMB/PZA
  Arms: Rifampicin group
Drug: Rifabutin — Rifabutin capsules, 150mg
  Other Names: Rifabutin/INH/EMB/PZA
  Arms: Rifabutin group

SUMMARY:
To compared the efficacy and safety of rifampicin and rifabutin which included in the standard treatment of anti-tuberculosis in HIV/AIDs patients combined with pulmonary tuberculosis, a multi-center, prospective cohort will be established. Antiviral efficacy and drug drug interaction will be investigated in order to provide optimized treatment for HIV/AIDs with tuberculosis.

DETAILED DESCRIPTION:
Two hundreds and thirty participants will be randomly assigned to receive an anti--tuberculosis treatment include rifampicin or rifabutin for two months of intensive therapy. Isoniazid and rifampicin (or rifabutin) will be continued to use for four months of consolidation therapy. A total of followed up period will be 12 months.

The antiretroviral therapy（ART） include:

Tenofovir disoproxil fumarate 300mg/d +Lamivudine 300mg/d+ Efavirenz 600mg/d; or Zidovudine 300mg bid +Lamivudine 300mg/d +Efavirenz 600mg/d.

ART will be started after 2 weeks of anti-tuberculosis.

The follow-up visits include 2th, 4th, 6th, 8th, 12th,16th, 20th, 24th, 32th, 36th, 40th, 44th and 48th week. sputum smear, sputum culture, chest X-ray, CD4 Lymphocyte counts,HIV viral load and adverse event will be tested and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years old;
2. No limited to gender;
3. If anti-HIV-1 positive samples are detected by an initial test based on the ELISA method, they should be confirmed by western blot;
4. The patients who are diagnosed with pulmonary TB (mycobacterium tuberculosis of sputum smear or culture was positive) but had never be treated;
5. Sign informed consent form voluntarily, and guarantee to attend follow-up visits;
6. Do not have plan to remove from the current experimental site during the trial process;
7. The patients do not receive any antiretroviral treatment before;
8. The overall situation of the patient should not affect the assessment and completion of the trial.

Exclusion Criteria:

1. Patients with acute infection;
2. During the screening period，patients with combined opportunistic infections and instability (National HIV/AIDS treatment guidelines) except for tuberculosis, or combined malignancy;
3. During the screening period，hemachrome < 6 g/dl, leukocyte < 2000 /µl, neutrophils < 1000 /µl, platelet count < 75000 /µl, blood amylase is greater than two times the upper limit of normal, Scr is greater than1.5 times the upper limit of normal, AST/ALT/AKP is greater than two times the upper limit of normal, TBIL is greater than two times the upper limit of normal, serum CK is greater than two times the upper limit of normal;
4. Now suffering from acute or chronic pancreatitis;
5. Now suffering from peripheral neuritis;
6. Pregnant and lactating women;
7. Patients with severe mental and neurological diseases;
8. Drug users；
9. Patients with history of heavy drinking and cannot be terminated;
10. Serious gastrointestinal ulcers；
11. Atherosclerosis affects the arteries in the heart, brain or kidneys；
12. Non-Chinese nationality；
13. Now suffering from myopathy；
14. Patients with previously treated tuberculosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of sputum negative conversion | 2~24 weeks
  The rate of the patients whose mycobacterium tuberculosis cannot be detected in sputum smear or bacteria culture.
Case fatality rate | 12 months
  The number of deaths during follow-up caused by HIV/AIDS and TB / the number of patients with HIV/AIDs and TB enrolled in this study * 100%.

SECONDARY OUTCOMES:
Treatment completion status | 12 months
  The rate of patients who complete the whole anti-tuberculous treatment.
The percentage of HIV viral load less than the detection limit | 6 months and 12 months
  The percentage of HIV viral load less than the detection limit
AE | 12 months
  The number and severity of adverse event.
Time of sputum negative conversion | 2~24 weeks
  The time of sputum negative conversion.
Chest CT scans improvement | 2~24 weeks
  Chest CT showed tuberculosis lesion absorption

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No